CLINICAL TRIAL: NCT07394491
Title: Intravenous Paracetamol Versus Intramuscular Tramadol in Shortening the Duration of Labour: a Randomized Controlled Trial
Brief Title: Intravenous Paracetamol Versus Intramuscular Tramadol in Shortening the Duration of Labour.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RE/M4H/86/22
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Labour Duration
Keywords: Labour duration; intramuscular tramadol; intravenous paracetamol
MeSH Terms: interventions — Acetaminophen; Tramadol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intramuscular tramadol (Active Comparator): 100mg of tramadol was given intramuscularly in active phase of labour
  Interventions: Drug: Tramadol hydrochloride
- paracetamol (Experimental): 1000mg of paracetamol given intravenously in active phase of labour
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: paracetamol — 1000 mg of paracetamol was administered intravenously to participants in active phase of labour
  Other Names: acetaminophen
  Arms: paracetamol
Drug: Tramadol hydrochloride — 100mg of tramadol given in active phase of labour
  Other Names: tramadol
  Arms: intramuscular tramadol

SUMMARY:
It is a well established fact that the pain of labour can be excrutiating and ways to shorten the duration of labour has been sought after. this study compares the role of intramuscular tramadol and intravenous paracetamol in shortening the duration of labour

DETAILED DESCRIPTION:
Background: The excruciating pain associated with labour as led to different studies aimed at finding pharmacolologic and non pharmacologic ways of shortening the duration of labour. Most agents used are either expensive or associated with fetomaternal adverse effects. This has led to the study of paracetamol and tramadol that have analgesic properties and have shown to have effect on labour duration.

Aim: To compare intravenous paracetamol versus intramuscular tramadol in shortening the duration of labour at Alex Ekwueme Federal University Teaching Hospital and St Patrick's Mile 4 Hospital, Abakaliki, Ebonyi State.

Methodology: It is an open label, non inferiority randomized controlled trial that was conducted on one hundred and eighty-nine parturients in active labour. Group A received 1000mg of intravenous paracetamol while Group B received 100mg of intramuscular tramadol and allocation was in the ratio of 1:1. Labour duration in the active phase was noted. Data were analyzed using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous active phase labour
* No contraindication to vaginal delivery

Exclusion Criteria:

* Clinical evidence of cephalopelvic disproportion
* Malpresentation,
* Multiple pregnancy,
* Previously scarred uterus,
* Preterm labour,
* Induced labour
* Antepartum hemorrhage.
* History of known allergy to tramadol and paracetamol or opioids or
* History of narcotics dependency.
* History of renal disease,
* Fetal distress
* Intrauterine fetal death.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Mean duration of first, second and third stage of labour | 12 hours
  the mean of the different stages of labour as well as the total duration of labour

CONTACTS AND LOCATIONS:
Overall Officials: Assumpta N Nweke, Principal Investigator — ST Patrick Mission Hospital, Mile $ Abakaliki, Ebonyi State
Locations (1):
- Assumpta Nnenna Nweke, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No